CLINICAL TRIAL: NCT01730729
Title: A Pilot Phase II Trial of Cabergoline in the Treatment of Metastatic Breast Cancer
Brief Title: Cabergoline in Metastatic Breast Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Lynn Sage Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 12B06; NCI-2012-02039 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STU00071477 (Other: Northwestern University IRB#)
Record Dates: First submitted 2012-11-15; First posted 2012-11-21 (Estimated); Results first posted 2019-03-26 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Recurrent Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cabergoline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (cabergoline) (Experimental): Patients receive cabergoline oral (PO) twice weekly for weeks 1-4. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cabergoline

INTERVENTIONS:
Drug: cabergoline — Given orally
  Other Names: Dostinex; FCE 21336

SUMMARY:
Prolactin is a hormone produced in the pituitary gland. Previous studies have revealed that elevated levels of the hormone prolactin might be associated with an increased risk of breast cancer. Cabergoline has been shown to lower prolactin levels in the blood.

The purpose of this study is to evaluate the effectiveness of cabergoline in treating metastatic breast cancer disease in those who test positive for the prolactin receptor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate overall response rate (ORR) of cabergoline in women with metastatic breast cancer.

SECONDARY OBJECTIVES:

I. Evaluate the progression-free survival (PFS) and overall survival (OS). II. Evaluate toxicity. III. Correlate serum prolactin levels during therapy with response. IV. Evaluate within-patient changes in computed tomography (CT) and bone scan measurements taken at baseline and after 2 cycles of treatment.

V. Evaluate within-patient changes in prolactin receptor (PRLr) expression from baseline to after 1 cycle of treatment in those patients who consent to optional repeat biopsy.

OUTLINE:

Patients receive cabergoline orally (PO) twice weekly for weeks 1-4. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed metastatic breast cancer; tissue (a minimum of 3 slides) from the most recent biopsy is required for review and confirmation of eligibility; NOTE: material should ideally be from the metastatic disease, however material from the primary tumor is acceptable if that is all that is available
* Patients must have stage IV breast cancer
* Patients must have tumors (primary or metastatic) that stain positively for the prolactin receptor
* Patients may have measurable or evaluable disease

  * Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as > 20 mm with conventional techniques or as > 10 mm with spiral CT scan
  * Evaluable disease is disease that does not meet the criteria for measurable disease; examples would include patients with effusions or bone-only disease
* Women of childbearing potential must commit to the use of effective barrier (non-hormonal) contraception while on study
* Patients must have a life expectancy of greater than 12 weeks
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Patients may have had a prior diagnosis of cancer if it has been > 5 years since their last treatment
* Leukocytes >= 3,000/uL (microliter)
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 100,000/uL
* Child Pugh score =< 10
* Patients must be able to swallow and retain oral medication
* All patients must have given signed, informed consent prior to registration on study

Exclusion Criteria:

* Women who are pregnant or lactating are not eligible for study treatment
* Patients who are undergoing concomitant radiotherapy are NOT eligible for participation
* Patients who are receiving any other investigational agents or concurrent anticancer therapy are NOT eligible for participation; previous systemic treatment is allowed with a 2 week washout period prior to registration
* Patients who are taking any herbal (alternative) medicines are NOT eligible for participation; patients must be off any such medications by the time of registration
* Patients who are receiving concomitant D2-antagonists (such as phenothiazines, butyrophenones, thioxanthenes, or metoclopramide) are NOT eligible for participation; patients must be off any such medications by the time of registration
* Patients with known brain metastases are NOT eligible for participation
* Patients with any of the following conditions or complications are NOT eligible for participation:

  * Uncontrolled hypertension
  * Known hypersensitivity to ergot derivatives
  * History of cardiac valvular disorders, as suggested by anatomical evidence of valvulopathy of any valve (to be determined by pre-treatment evaluation including echocardiographic demonstration of valve leaflet thickening, valve restriction, or mixed valve restriction-stenosis)
  * History of pulmonary, pericardial, cardiac valvular, or retroperitoneal fibrotic disorders
  * Gastrointestinal (GI) tract disease resulting in an inability to take oral medication
  * Malabsorption syndrome
  * Require intravenous (IV) alimentation
  * History of prior surgical procedures affecting absorption
  * Uncontrolled inflammatory GI disease (e.g., Crohn's, ulcerative colitis)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-02-11 (Actual); Primary Completion 2015-12-15 (Actual); Study Completion 2017-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Kaklamani, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened for accrual on November 29, 2012 with an accrual goal of up to 20 patients. The first patient starting treatment February 11, 2013. Accrual was suspended twice during the study; May 28 2014 reopening June 11, 2014 and July 24 2015, reopening August 27 2015. The study was closed October 21, 2015 with 20 patients enrolled.
Period: Overall Study
Arm/Group | Treatment (Cabergoline)
Started | 20
Completed 2 Cycles/Reached 1st Response | 18
Treated Cycle 3 and Beyond | 6
Completed (Patients treated until progressive disease, unacceptable toxicity, or withdrawal from study) | 6
Not Completed | 14
Not completed — Adverse Event | 1
Not completed — Death | 1
Not completed — Progressive Disease | 12

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Cabergoline)
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) at 2 Months
Description: Overall Response Rate (ORR) is defined as the number of patients that achieved Complete Response (CR) or Partial Response (PR) and will be assessed after 8 weeks (2 cycles) of therapy using CT scan images and RECIST guidelines.
  Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum of LD.
  Progressive Disease (PD): At least a 20% increase in the sum o the LD of target lesions, taking as reference the smallest sum of LD recorded since the treatment started or the appearance of one or more new lesions.
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of LD since the treatment started
Time Frame: After 8 weeks (2 cycles) of treament
Population: 2 patients did not reach 8 week response time point and were determined not to be evaluable for this objective.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Cabergoline)
Number analyzed (Participants) | 18
Participants | 0

2. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression Free Survival (PFS) will be measured from time of treatment initiation until first documentation of progression of disease or death from any cause.
Time Frame: From start of treatment until progression of disease or death
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Cabergoline)
Number analyzed (Participants) | 20
Months | 1.84 [1.84 to 3.68]

3. Secondary Outcome: Treatment Toxicity
Description: Toxicity will be assessed at the beginning of each cycle (1 cycle equals 28 days) during treatment and 30 days post last treatment during treatment. Toxicity will be assessed according to the National Cancer Institute's Common Toxicity Criteria for adverse events version 3.0 (CTCAE v3.0). In general adverse events (AEs) will be graded according to the following:
  Grade 1 Mild AE Grade 2 Moderate AE Grade 3 Severe AE Grade 4 Life-threatening or disabling AE Grade 5 Death related to AE Grades 1 through 4 adverse events that were determined to be at least possibly related to treatment are combined and reported below.
Time Frame: After every 4 weeks (1 cycle) during treatment for up to 20 cycles and 30 days post last treatment
Measure: Number; unit: participants
Arm/Group | Treatment (Cabergoline)
Number analyzed (Participants) | 20
participants
  Nausea | 6
  Fatigue | 5
  Hyponatremia | 3
  Alkaline Phosphatase increased | 3
  Aspartate Aminotansferase increased | 2
  Hyperglycemia | 2
  Hypokalemia | 2
  Vomiting | 1
  Pain in extremity | 1
  Acute Kidney Injury | 1
  Alanine Aminotranserase increased | 1
  Arthralgia | 1
  Creatinine increased | 1
  Diarrhea | 1
  Dizziness | 1
  Dry eye | 1
  Hyperkalemia | 1
  Hypernatremia | 1
  Hypocalcemia | 1
  Hypoglycemia | 1
  Insomnia | 1
  Pain | 1
  White Blood Cell decreased | 1

4. Secondary Outcome: Change in Within-patient Imaging Measurements at Baseline and After 2 Cycles
Description: At baseline and after 2 cycles changes CT and bone scan measurements will be evaluated.
Time Frame: At baseline and at 8 weeks
Population: This data was not collected and analysed as it was decided that it was not meaningful on its own.
Arm/Group | Treatment (Cabergoline)
Number analyzed (Participants) | 0

5. Secondary Outcome: Change in Prolactin Receptor Expression Measurements at Baseline and After 1 Cycle
Description: Evaluate prolactin expression in biopsy tissue taken at baseline and after 4 weeks (1 cycle) of treatment.
Time Frame: At baseline and after 4 weeks (1 cycle)
Population: No data collected as no patients completed repeat biopsy after 1 cycle of treatment.
Arm/Group | Treatment (Cabergoline)
Number analyzed (Participants) | 0

6. Secondary Outcome: Correlate Tissue Prolactin Biomarkers With Response to Therapy
Description: Baseline tumor tissue was analyzed for prolactin receptor (PRLr) expression and was provided with an IHC-based Allred score of 0 to 300 based on percentage intensity where lower scores indicate less PRLr expression and high scores indicate more PRLr expression. Only the malignant epithelium was scored. The score was correlated with best response of patient.
Time Frame: At baseline
Population: Only 9 patients had sufficient baseline tissue to be analyzed.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Treatment (Cabergoline)
Number analyzed (Participants) | 9
score on a scale
  Stable Disease: number analyzed (Participants) | 3
  Stable Disease | 170 [110 to 220]
  Progressive Disease: number analyzed (Participants) | 6
  Progressive Disease | 220 [120 to 250]

7. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) is defined from the first day of treatment until death from any cause.
Time Frame: From the start of treatment until death from any cause. Median follow up time of 6.817 months (95%CI 0.22-26.18)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Cabergoline)
Number analyzed (Participants) | 20
Months | 10.41 [7.06 to NA] — At the time of data collection cut off, not all patients were deceased and upper CI was not calculated.

8. Post Hoc Outcome: Clinical Benefit Rate (CBR) After 2 Cycles of Treatment
Description: Clinical Benefit Rate (CBR) is defined as the number of patients with Complete Response (CR), Partial Response (PR), or Stable Disease (SD) and is assessed by RECIST guidelines for measurements of CT scan at 8 weeks (2 cycles) of treatment.
  Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum of LD.
  Progressive Disease (PD): At least a 20% increase in the sum o the LD of target lesions, taking as reference the smallest sum of LD recorded since the treatment started or the appearance of one or more new lesions.
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of LD since the treatment started
Time Frame: After 8 weeks (2 cycles) of treatment
Population: 2 patients did not reach the 8 week response assessment time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Cabergoline)
Number analyzed (Participants) | 18
Participants | 6

9. Post Hoc Outcome: Disease Control at 12 Months
Description: Number of patients without progressive disease as assessed by CT scan and RECIST guidelines at 12 months of treatment.
Time Frame: At 12 months from start of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Cabergoline)
Number analyzed (Participants) | 20
Participants | 2

10. Post Hoc Outcome: Best Overall Response
Description: Best Overall Response is defined as patients best response to treatment from treatment initiation until the end of treatment as assessed by RECIST guidelines of CT scans.
  Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum of LD.
  Progressive Disease (PD): At least a 20% increase in the sum o the LD of target lesions, taking as reference the smallest sum of LD recorded since the treatment started or the appearance of one or more new lesions.
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of LD since the treatment started
Time Frame: From the start of treatment until the end of treatment up to a maximum of 20 cycles (1 cycle = 4 weeks)
Population: 1 patient died on treatment 7 days after starting and was not included in this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Cabergoline)
Number analyzed (Participants) | 19
Participants
  Partial Response | 1
  Stable Disease | 5
  Progressive Disease | 13

11. Post Hoc Outcome: Change in Serum Prolactin Levels From Baseline and After 2 Cycles of Treatment
Description: Serum prolactin measurements were taken at baseline and after completion of two cycles of treatment. The mean drop was calculated for all patients, and for patients with best response of Stable Disease and Progressive Disease.
Time Frame: At baseline and after 2 cycles of treatment where 1 cycle =4 weeks
Population: Serum prolactin at baseline and after 2 cycles of treatment were only available for 12 patients.
Measure: Mean (Full Range); unit: ng/ml
Arm/Group | Treatment (Cabergoline)
Number analyzed (Participants) | 12
ng/ml
  All | -9.425 [-36.70 to -0.50]
  Stable Disease: number analyzed (Participants) | 5
  Stable Disease | -8.72 [-11.50 to -5.50]
  Progressive Disease | -9.93 [-36.70 to -0.50]

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a 3 year period for the whole study. Patients were followed from treatment initiation, throughout treatment and 30 days post last treatment for up to 20 cycles (max number of cycles that any patient was treated) where 1 cycle equals 28 days.
Arm/Group | Treatment (Cabergoline)
All-Cause Mortality (participants affected / at risk) | 13/20
Serious Adverse Events (participants affected / at risk) | 4/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Cabergoline) (N=20)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Death NOS (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Cabergoline) (N=20)
Anemia (Hemoglobin decrease) (Blood and lymphatic system disorders) | 6
Sinus Tachycardia (Cardiac disorders) | 2
Dry eye (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Oral Mucositis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 6
Stomach pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Edema limbs (General disorders) | 1
Fatigue (General disorders) | 7
Alanine aminotransferase increased (Investigations) | 2
Alkaline phosphatase increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 13
Blood prolactin abnormal (Investigations) | 15
Cardiac troponin 1 increased (Investigations) | 1
Creatinine increased (Investigations) | 2
INR increased (Investigations) | 1
Lymphocyte Count decreased (Investigations) | 10
Platelet Count decreased (Investigations) | 2
Weight loss (Investigations) | 1
White Blood Cell decreased (Investigations) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 12
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 9
Hypocalcemia (Metabolism and nutrition disorders) | 7
Hypoglycemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Investigations) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Headaches (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Acute Kidney Injury (Renal and urinary disorders) | 1 — Low grade - Not resulting in hospitalization
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 1
Erythematous papules (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1
Lymphedema (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No